CLINICAL TRIAL: NCT06844279
Title: Geriatrik Hasta Grubunda Anestezi Derinliği Monitörizasyonlarının Postoperatif Derlenme ve Bilişsel Fonksiyonlara Etkileri
Brief Title: The Effects of Anesthesia Depth Monitoring on Postoperative Recovery and Cognitive Functions in the Geriatric Patient Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aslıhan Güleç (Other)
Responsible Party: Sponsor-Investigator, Aslıhan Güleç, MD, Specialist in Anesthesiology and Reanimation, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Gazi-2024 -1816
Record Dates: First submitted 2025-02-09; First posted 2025-02-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Geriatric Patient Care Improvement; Postoperative Delirium (POD); Burst Suppression
Keywords: anaesthesia depth monitoring; geriatric; density spectral array; bispectral index; burst supression; postoperative delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Group 1: Anaesthesia depth monitoring according to hemodynamic values Group 2: Anaesthesia depth monitoring according to numeric BIS values (numbers between 40 to 60 is aimed) Group 3: Anaesthesia depth monitoring according to DSA function (avoiding obvious burst supression and keeping alpha band in high frequency)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Hemodynamic-Guided Group (Active Comparator): Anesthesia depth monitoring will be managed according to hemodynamic parameters, primarily avoiding hypotension.
  Interventions: Other: Control Group: Standard Hemodynamic Monitoring
- BIS-Guided Group (Active Comparator): Anaesthesia depth monitoring according to numeric BIS index values
  Interventions: Device: Processed Electroencephalogram (BIS Index)
- DSA-Guided Group (Active Comparator): Anesthesia depth monitoring using the Density Spectral Array (DSA) function of the BIS monitor.
  Interventions: Device: Processed Electroencephalogram (DSA Mode)

INTERVENTIONS:
Other: Control Group: Standard Hemodynamic Monitoring — Anesthesia depth monitoring based on hemodynamic values without additional processed EEG guidance.
  Arms: Hemodynamic-Guided Group
Device: Processed Electroencephalogram (BIS Index) — Anaesthesia depth monitoring according to numeric BIS index values.
  Arms: BIS-Guided Group
Device: Processed Electroencephalogram (DSA Mode) — Anaesthesia depth monitoring according to density spectral array functions
  Arms: DSA-Guided Group

SUMMARY:
This study will be conducted on patients aged 65 and older scheduled for surgery due to lumbar or cervical disc herniation. General anesthesia is routinely used for these types of surgeries in the hospital. In patients receiving general anesthesia, anesthesia depth monitoring is performed.

As part of the study, a preoperative anesthesia evaluation will be conducted, which will include age, weight, height, comorbidities, regularly used medications, previous surgical or anesthesia experiences, nutritional habits, mental status, and daily activity levels.

On the day of surgery, upon arrival in the operating room, the following will be measured and recorded:

* Blood pressure using a non-invasive blood pressure monitor
* Heart rate and rhythm via electrocardiogram (ECG)
* Blood oxygen level with a pulse oximeter
* Anesthesia depth using a forehead-applied sensor

All monitoring procedures are non-invasive and painless. Following the placement of these monitoring devices and initial measurements, anesthesia induction and surgery will commence. Throughout surgery, blood pressure, heart rate, and brain activity will be continuously recorded. After the surgical procedure, anesthesia emergence and mental status will be assessed. Preoperative evaluation data and intraoperative recordings will be used solely for research purposes, with patient identity information remaining confidential.

DETAILED DESCRIPTION:
Perioperative cognitive decline and delirium occur more frequently in the geriatric population undergoing surgery. International guidelines recommend monitoring anesthesia depth to reduce the risk of postoperative cognitive dysfunction. Anesthesia depth is commonly measured using non-invasive electroencephalography (EEG)-based methods, such as the Bispectral Index (BIS).

Previous studies have predominantly utilized processed EEG monitors that generate numerical values for tracking anesthesia depth. However, in this study, anesthesia depth will be monitored using both the standard numerical BIS index and the Density Spectral Array (DSA) mode, an advanced feature of the BIS device. To date, no studies have simultaneously examined BIS and DSA modes in relation to cognitive function and the recovery process.

The use of advanced monitoring techniques may serve as a valuable resource for future research, particularly in optimizing anesthetic management for geriatric patients with reduced cognitive reserve. This study aims to evaluate the effects of different intraoperative anesthesia depth monitoring approaches, including hemodynamic monitoring, numerical BIS values, and DSA functions. The primary objective is to determine the optimal anesthesia monitoring strategy that minimizes intraoperative hypotension, burst suppression, and postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Elective spinal surgeries
* ASA status I-III

Exclusion Criteria:

* Emergent surgeries
* ASA status IV-V
* Prediagnosed delirium and or dementia
* Inability to give consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Ratio of Burst Suppression | Intraoperative (continuously recorded from anesthesia induction to emergence)
  The burst suppression ratio (BSR) will be calculated as the percentage of total anesthesia time spent in burst suppression, as measured by processed electroencephalography (EEG). A higher BSR has been associated with worse postoperative cognitive outcomes.
Time of Burst Suppression | Intraoperative (continuously recorded from anesthesia induction to emergence)
  Anesthesia time spent in burst suppression (BS), as measured by processed electroencephalography (EEG). A higher BS time has been associated with worse postoperative cognitive outcomes.
Intraoperative Hypotension Incidence | Intraoperative (assessed continuously throughout surgery)
  Intraoperative hypotension will be measured in 5-minute intervals. Hypotension is a mean arterial pressure (MAP) below 60 mmHg. The episodes of hypotension at any point during surgery will be recorded.
Alpha Band Preservation or Loss | Intraoperative (measured continuously from anesthesia induction to emergence)
  Alpha band activity (8-12 Hz) in the frontal lobe will be evaluated to determine whether it is preserved or lost during general anesthesia. Alpha band preservation is associated with optimal anesthesia depth and cognitive function preservation, while loss of alpha band activity is linked to increased postoperative cognitive impairment.

SECONDARY OUTCOMES:
Incidence of Postoperative Delirium Assessed via CAM Scale | Postoperative (assessed at 6, 24, and 48 hours after surgery)
  Postoperative delirium will be assessed using the Confusion Assessment Method (CAM) tool. The number of participants meeting the criteria for delirium within the first 48 hours postoperatively will be recorded.
Total Intraoperative Propofol Consumption | Intraoperative
  The total dose of propofol administered intraoperatively will be recorded. Data will be reported as mg/kg.
Total Intraoperative Sevoflurane Consumption | Intraoperative
  The total dose of Sevoflurane administered intraoperatively will be recorded. Data will be reported as ml.
Total Intraoperative Remifentanil Consumption | Intraoperative
  The total dose of Remifentanil administered intraoperatively will be recorded. Data will be reported as mcg/kg.
Total Intraoperative Vasopressor Consumption | Intraoperative
  The total dose of vasopressors (noradrenaline, adrenaline, dopamine) administered intraoperatively will be recorded. Data will be reported as mcg/kg.

OTHER OUTCOMES:
Frailty Score Assessed via Clinical Frailty Scale (CFS) | Preoperative (assessed on the day of surgery)
  Frailty will be assessed preoperatively using the Clinical Frailty Scale (CFS), which ranges from 1 (very fit) to 9 (terminally ill). Higher scores indicate worse frailty status. The proportion of participants classified as frail (CFS ≥ 5) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Zerrin Ozkose Satirlar, Professor, Study Director — Gazi University
Locations (1):
- Gazi University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in the publication
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending one year after the publication
Access Criteria: Access to study protocol upon request, contact with one of the sub-investigators.

REFERENCES:
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Wildes TS, Mickle AM, Ben Abdallah A, Maybrier HR, Oberhaus J, Budelier TP, Kronzer A, McKinnon SL, Park D, Torres BA, Graetz TJ, Emmert DA, Palanca BJ, Goswami S, Jordan K, Lin N, Fritz BA, Stevens TW, Jacobsohn E, Schmitt EM, Inouye SK, Stark S, Lenze EJ, Avidan MS; ENGAGES Research Group. Effect of Electroencephalography-Guided Anesthetic Administration on Postoperative Delirium Among Older Adults Undergoing Major Surgery: The ENGAGES Randomized Clinical Trial. JAMA. 2019 Feb 5;321(5):473-483. doi: 10.1001/jama.2018.22005. PMID 30721296
- [Background] Chen YC, Hung IY, Hung KC, Chang YJ, Chu CC, Chen JY, Ho CH, Yu CH. Incidence change of postoperative delirium after implementation of processed electroencephalography monitoring during surgery: a retrospective evaluation study. BMC Anesthesiol. 2023 Oct 4;23(1):330. doi: 10.1186/s12871-023-02293-9. PMID 37794315
- [Background] Shao YR, Kahali P, Houle TT, Deng H, Colvin C, Dickerson BC, Brown EN, Purdon PL. Low Frontal Alpha Power Is Associated With the Propensity for Burst Suppression: An Electroencephalogram Phenotype for a "Vulnerable Brain". Anesth Analg. 2020 Nov;131(5):1529-1539. doi: 10.1213/ANE.0000000000004781. PMID 33079876
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878